CLINICAL TRIAL: NCT06654895
Title: Multicenter Symphony IL-6 Monitoring Sepsis ICU Validation Study
Acronym: SYMON II
Status: Recruiting | Type: Observational
Sponsor: Bluejay Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CES-0008
Record Dates: First submitted 2024-10-15; First posted 2024-10-23 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-12

CONDITIONS: Sepsis, Septic Shock
Keywords: Interleukin-6; IL-6; Risk Stratification; Infections; Toxima; Systemic Inflammatory Response Syndrome; Inflammation; Pathologic Processes; Sepsis; Septic Shock; Shock
MeSH Terms: conditions — Sepsis; Shock, Septic; Infections; Systemic Inflammatory Response Syndrome; Inflammation; Pathologic Processes; Shock

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of this study is to validate a pre-defined IL-6 concentration cutoff that predicts 28-day mortality in patients who are admitted or are intended to be admitted to the ICU diagnosed with sepsis or septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥22 years of age)
* Diagnosis of sepsis or septic shock based on: the Third International Consensus Definitions (Sepsis-3 criteria) defined as at least one of the following criteria as determined by a treating physician or study physician investigator.

  * Sepsis: suspected or documented infection (i.e., use or intent to use antibiotics as an indicator) and organ dysfunction defined by a Sequential Organ Failure Assessment (SOFA) score ≥2
  * Septic shock: sepsis requiring vasopressors and serum lactate levels >2 mmol/L (18 mg/dL)
* Admitted or intended to be admitted to the ICU
* At least 3 mL plasma drawn and available for collection (or is anticipated to be able to be drawn and available) within 24 hours of (i.e., up to 24 hours after) the earliest diagnosis of sepsis or septic shock.

Exclusion Criteria:

* Prisoners or imprisonment at time of enrollment
* Prior enrollment into this study
* Informed consent as approved by IRB is unable to be obtained.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with sepsis or septic shock, in accordance with the sepsis-3 criteria, admitted or intended to be admitted to the ICU.
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
28-day all-cause mortality [Time Frame: within 28 days after inclusion] participants will be followed up for 28 days | Within 28 days after inclusion
  Participants will be followed up for 28 days for all-cause mortality

SECONDARY OUTCOMES:
In-hospital mortality up to 28 days | Within 28 days after inclusion
  Participants will be followed up for 28 days for in-hospital mortality
All-cause mortality up to 7 days | Within 7 days after inclusion
  Participants will be followed up for 7 days for all-cause mortality
Sequential Organ Failure Assessment (SOFA) score | Within 28 days after inclusion
  SOFA score has a range from 1 to 24, where higher scores represent higher degrees of single or multiple organ failure(s).
Hospital length of stay | Within 28 days after inclusion
  Participants will be followed up for hospital length of stay for up to 28 days
ICU length of stay | Within 28 days after inclusion
  Participants will be followed up for ICU length of stay for up to 28 days
Vasopressor utilization | Within 28 days after inclusion
  Participants will be followed up for use of Vasopressors for up to 28 days
Progression to septic shock | Within 28 days after inclusion
  Participants will be followed up for progression to septic shock for up to 28 days
28-day all-cause mortality in patients with a final diagnosis of sepsis or septic shock | Within 28 days after inclusion
  Participants will be followed up for 28 days for all-cause mortality

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of Florida College of Medicine, Gainesville, Florida
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Wake Forest School of Medicine, Winston-Salem, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Intermountain Health, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No